CLINICAL TRIAL: NCT04442256
Title: Effect of Dupilumab on ASS Intolerance and Its Mechanisms in Patients With Aspirin-exacerbated Respiratory Disease (AERD)
Brief Title: Effect of Dupilumab on Aspirin Intolerance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Tamara Quint, Principal investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004889-18
Record Dates: First submitted 2020-06-03; First posted 2020-06-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: AERD - Aspirin Exacerbated Respiratory Disease
Keywords: AERD; Asthma; Morbus Widal; chronic rhinosinusitis with nasal polyps; dupilumab
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Only one group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupilumab (Other): All patients will be administered subcutaneous doses of dupilumab in a monthly fashion. Observation period will be 30 minutes after injection
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — All patients will be administered subcutaneous doses of dupilumab in a biweekly fashion.

SUMMARY:
To test the efficacy of dupilumab in patients with AERD regarding the intolerance to salicylic acid after 6 months. This will be evaluated by oral drug provocation testing with low dose salicylic acid after 6 months of dupilumab treatment.

Hypothesis:

After 6 months of therapy, patients will tolerate aspirin dose levels as tested with different dosages (125mg, 250mg and 500 mg).

DETAILED DESCRIPTION:
30 patients suffering from AERD will be included in this single-center, prospective, explorative study for treatment with dupilumab. Before study initiation, informed consent will be obtained from all subjects. All patients with AERD can be included according to inclusion- and exclusion criteria.

AERD patients who had already obtained a monoclonal antibody for the treatment of asthma or polyps will also be included if at least a wash out period of 5 half -lives or 3 months has passed. The first visit will be performed at screening (day 0, V1/before dupilumab therapy). Clinically significant abnormal laboratory values will be ruled out prior to the first dose.

All patients will be administered subcutaneous doses of dupilumab in a biweekly fashion.

For several reasons comparison with placebo will not be performed:

* All patients included are in urgent need for an effective treatment.
* The only currently available alternative treatment option is a functional endoscopic sinus surgery (FESS). Usually there is a high recurrence rate after surgery.
* All included patients have a long medical history concerning AERD. The rate of a spontaneous improvement or resolution in this patient population is negligible.

Spirometry (peak-flow and FEV1) and an asthma control test will be performed prior to dupilumab therapy, after 1, 3 and 6 months. In addition, the sinonasal outcome test-22 and the total nasal endoscopic polyps score as well as nasal congestion score, disease severity (by visual analogue scale=VAS), total symptom score (TSS) will be performed at baseline, after 1,3 and 6 months. To further evaluate the polyp size, a nasal CT will be performed at screening visit. To evaluate the sense of smell we will perform UPSIT testing before and after 6 months dupilumab.

All patients will have routine laboratory testing (blood chemistry, hematology) before and after 6 months of therapy. Adverse events will be recorded at each visit. Biological activity will be evaluated based on peripheral blood eosinophil counts, serum total Immunoglobulin E (IgE) levels and measurement of eosinophilic cationic protein in patients' sera at baseline and after 6 months.

To assess local changes in the nose caused by dupilumab treatment, nasal secretions, nasal mucosa samples (nasal curette), nasal microbiome as well as nasal biopsies will be collected.

After the end of study, treatment will be continued in all patients with significant improvement in asthmatic symptoms, nasal symptoms as well as a reduction of polyps.

For patients who did not experience clinical improvement, dupilumab treatment will be discontinued after 6 months.

ELIGIBILITY:
Inclusion Criteria:

Dupilumab treatment group:

* Signed and dated informed consent has been obtained
* Age 18 - 70 years
* Male or female
* Diagnosed with AERD (nasal polyps, allergic asthma, aspirin intolerance)
* Chronic rhinosinusitis with nasal polyps (CRSwNP) (according to the European Position Paper on Rhinosinusitis and Nasal Polyps Guidelines)8
* Documented aspirin intolerance
* Asthma bronchial diagnosed by a respiratory physician (based on Global -Initiative for Asthma guidelines)9

Exclusion Criteria:

* Pregnancy
* Clinically significant abnormal laboratory values and active infection (Tbc, HIV, hepatitis A/B/C)
* History of malignancy or immunodeficiency
* Chronic obstructive lung disorders (COPD), other obstructive lung disorders (bronchiolitis)
* Need for systemic corticosteroid therapy 1 month prior to screening visit Eosinophilic pneumonia and Churg-Strauss Syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated aspirin dose level (stages 125mg, 250mg and 500mg) | 6 months
  Changes in the maximal ASS dose level tolerations (no toleration, 125mg, 250mg and 500mg) at baseline and after 6 months.

SECONDARY OUTCOMES:
Change of nasal polyps (TPS) | 6 months
  A secondary endpoint is the change of polyps after 6 months of treatment with dupilumab, which will be evaluated by an ENT specialist. The polyps will be evaluated on each side by means of nasal endoscopy and graded based on polyp size, resulting in scores of 0 to 4 (TPSs).
Change of allergic asthma (Spirometry) | 6 months
  Changes in spirometry (FEV1%)
Percentage of T and B cell subsets in nasal polyp tissues of patients treated with dupilumab as assessed with confocal microscopy | 6 months
  Biopisies of nasal polyps will be taken at baseline and after 6 months of treatment with Dupilumab. RNA will be isolated from part of the biopsy and subjected to bulk RNA sequencing. Genes up or downregulated upon treatment will be calculated by bioinformaticians. Biopsies will also be assessed by confocal microscopy upon staining for surface specific markers identifiying various T (T mem, reg T cells) and B (Plasma cell, memory cells) as well as other immune cell subpopulations.
Change of allergic asthma (Asthma control test) | 6 months
  Change from baseline in allergic asthma on the asthma control test at 6 months.
Change of nasal polyps (SNOT-22) | 6 months
  Changes in sinus nasal outcome test-22 (SNOT 22) between baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bangert, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Eckl-Dorna J, Morgenstern C, Poglitsch K, Arnoldner T, Gangl K, Bartosik TJ, Campion NJ, Tu A, Stanek V, Schneider S, Bangert C. Dupilumab Dampens Mucosal Type 2 Response During Acetylsalicylic Acid Challenge in N-ERD Patients. Clin Exp Allergy. 2025 Nov 27. doi: 10.1111/cea.70184. Online ahead of print. PMID 41309110